CLINICAL TRIAL: NCT06289088
Title: The Effect of an Individually Adapted Lumbosacral Orthosis on Plantar Pressure and Balance in Individuals With Low Back Pain
Brief Title: The Effect of an Individually Adapted Lumbosacral Orthosis on Plantar Pressure and Balance
Acronym: lumbosacral
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve yilmaz menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: E-10840098-772.02-4659
Record Dates: First submitted 2024-02-26; First posted 2024-03-01 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Orthosis; Low Back Pain, Postural
Keywords: Low back pain; lumbosacral orthosis; orthosis adjustment; postural control; plantar pressure; balance
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Single group, crossover study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First Intervention (Experimental): The application will be done sequentially: without orthosis, with adaptation and with orthosis.
  Interventions: Other: First Intervention
- Second Intervention (Experimental): The application will be done sequentially: with adaptation, with orthosis and without orthosis
  Interventions: Other: Second Intervention
- Third Intervention (Experimental): The application will be done sequentially: with orthosis, without orthosis, and with adaptation
  Interventions: Other: Third Intervention

INTERVENTIONS:
Other: First Intervention — Firstly, For individuals with low back pain, all measurements will be evaluated without wearing any orthosis. The waist circumference of individuals with low back pain will be measured and the orthosis was adapted to the appropriate orthosis size by the prosthetist orthotist. After waiting with the orthosis for half an hour, the measurements will be repeated. Then, the person will be asked to wear the orthosis without any intervention.
  Arms: First Intervention
Other: Second Intervention — Firstly, The waist circumference of individuals with low back pain will be measured and the orthosis will be adapted to the appropriate orthosis size by the prosthetist orthotist. After waiting with the orthosis for half an hour, the person will be asked to wear the orthosis without any intervention and the outcome measurements will be repeated. After waiting with the orthosis for half an hour, all measurements will be evaluated without wearing any orthosis.
  Arms: Second Intervention
Other: Third Intervention — Firstly, the person will be asked to wear the orthosis without any intervention and the outcome measurements will be done. The waist circumference of individuals with low back pain will be measured and the orthosis will be adapted to the appropriate orthosis size by the prosthetist orthotist. After waiting with the orthosis for half an hour, all measurements will be evaluated without wearing any orthosis. Lastly, The waist circumference of individuals with low back pain will be measured and the orthosis will be adapted to the appropriate orthosis size by the prosthetist orthotis. After waiting with the orthosis for half an hour, all measurements will be evaluated.
  Arms: Third Intervention

SUMMARY:
The aim of this study is to examine the effect of steel underwire lumbosacral orthosis adapted to the individual by the prosthetist orthotist on pain, comfort, plantar pressure, static and dynamic balance in individuals with low back pain.

DETAILED DESCRIPTION:
The aim of this study is to examine the effect of steel underwire lumbosacral orthosis adapted to the individual by the prosthetist orthotist on pain, comfort, plantar pressure, static and dynamic balance in individuals with low back pain. Thirty male and female volunteers between the ages of 18-65 who came to Istanbul Medipol University Prosthesis Orthotics Center and experienced low back pain were included in the study.

The study will be designed as Crossover. The study consists of three methods and a single group, which are orthosis-free, worn by a person with low back pain, and adapted by a prosthetist orthotist. Following both orthosis insertion methods, pain severity will be measured with Visual Analogue Scale (VAS) and comfort level was measured with Orthosis Comfort Score. They will be asked to wait for 30 minutes with orthosis, and then the pain severity and comfort level were measured again. Y Balance Test (YBT) and Functional Reach Test (FRT) will be used for dynamic balance. Plantar pressure and static balance will be analyzed with pedobarography device. Static Pressure and stabilometric data will be found.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65,
* One or more recurrent low back pain during the last 12 months,-At least 6 points on the Oswestry Disability Index,
* Negative straight leg raising test result,
* Not having any lower extremity injuries in the last 6 months,
* No history of recent trauma or infection

Exclusion Criteria:

* Neurological symptoms due to nerve root compression
* One-sided leg pain more severe than lower back pain, pain in feet and toes shooting pain, numbness in the same area, paresthesia,
* Disease that causes neurological sequelae (stroke, traumatic brain injury, Parkinson's, Those who have had it (such as multiple sclerosis),
* Presence of malignancy,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-05-04 (Estimated); Study Completion 2024-05-04 (Estimated)

PRIMARY OUTCOMES:
Visual Analog scale | 5 minutes
  A Visual Analogue Scale (VAS) is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson[1]. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. For example, the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. From the patient's perspective, this spectrum appears continuous; their pain does not take discrete jumps, as a categorization of none, mild, moderate and severe would suggest. It was to capture this idea of an underlying continuum that the VAS was devised
Orthosis comfort score | 10 minutes
  An orthosis comfort score, which is valid and reliable and developed from the socket comfort score, will be used to evaluate comfort. The score measures the comfort felt by the patient between values of 0 and 10. "How would you rate the comfort of the orthosis?" They are expected to answer the question as 0 is the most uncomfortable orthosis and 10 is the most comfortable orthosis.
Functional Reach Test (FRT) | 5 minutes
  Functional Reach Test (FRT) is a assessment tool for ascertaining dynamic balance in in simple task. In standing, measures the distance between the length of an outstretched arm in a maximal forward reach, while maintaining a fixed base of support. This information is correlated with risk of falling.
Pedobarographic evaluation | 5 minutes
  Foot plantar pressure distribution (static pedobarographic) analyzes and postural stability parameters will be performed through a computer-aided data collection and display system. Sensor Medica (Rome, Italy) Pedobarography Device, which has a pressure-sensitive platform connected to the computer and a software system that records and analyzes the data. Measurements will be made for individuals with low back pain.
Y balance test | 15 minutes
  Y Balance Test, strength, flexibility, filter control and proprioception.Taking a one-legged stand is a reliable test for exercising dynamic balance. Three-way reach carries out operations of individuals of individuals. They were asked to lie down to the last magnification without disrupting the alignment with the side to be tested and to return to the center after each stretch. After trial access, access was requested in three directions. Measurements are fired with 10-second breaks between trials and 20-second breaks between directions. The reach made after 3 reach attempts for each direction was measured and taken into the recording area, and the test was used in the overall performance analysis.

CONTACTS AND LOCATIONS:
Overall Officials: MERVE YILMAZ MENEK, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Result] Azadinia F, Ebrahimi-Takamjani I, Kamyab M, Asgari M, Parnianpour M. Immediate Effects of Lumbosacral Orthosis on Postural Stability in Patients with Low Back Pain: A Preliminary Study. Arch Bone Jt Surg. 2019 Jul;7(4):360-366. PMID 31448314
- See also: Immediate Effects of Lumbosacral Orthosis on Postural Stability in Patients with Low Back Pain: A Preliminary Study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6686069/pdf/ABJS-7-360.pdf